CLINICAL TRIAL: NCT05315258
Title: A Phase II Non-Randomized, Open-label, Multi-centre Study of the Safety and Efficacy of Tebentafusp in Melanoma With Molecular Relapsed Disease
Brief Title: Tebentafusp in Molecular Relapsed Disease (MRD) Melanoma
Acronym: TebeMRD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTO_101; 2019-003946-34 (EudraCT Number)
Record Dates: First submitted 2021-08-23; First posted 2022-04-07 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Melanoma (Skin); Melanoma, Uveal
Keywords: D008545
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cutaneous melanoma with molecular relapsed disease (Experimental): tebentafusp weekly IV escalating in the first treatment cycle with dose 20 mcg on day 1, 30 mcg on day 8, 68 mcg on days 15 and 22. Thereafter weekly doses will be 68 mcg IV for 6 months.
  Interventions: Drug: Tebentafusp
- Uveal melanoma with molecular relapsed disease (Experimental): tebentafusp weekly IV escalating in the first treatment cycle with dose 20 mcg on day 1, 30 mcg on day 8, 68 mcg on days 15 and 22. Thereafter weekly doses will be 68 mcg IV for 6 months.
  Interventions: Drug: Tebentafusp

INTERVENTIONS:
Drug: Tebentafusp — Tebentafusp supplied as concentrate for solution for infusion and diluted prior to administration. 0.2 mg/mL drug product will be provided as a sterile, refrigerated solution in glass vials.
  Other Names: IMCgp100

SUMMARY:
Researchers are trying to find ways to improve the management of people with intermediate or high risk resected cutaneous melanoma or with primary uveal melanoma.

This research study is investigating using a new blood test to decide when to give a drug called tebentafusp. Tebentafusp has been used in clinical trials in patients with advanced cutaneous and uveal melanoma. This study is designed to determine if tebentafusp can help patients with cutaneous or uveal melanoma live longer.

DETAILED DESCRIPTION:
TebeMRD is an unblinded non-randomised, open labelled, safety and efficacy study involving 2 patient cohorts:

* A: Cutaneous melanoma with molecular relapsed disease (MRD)
* B: Uveal melanoma with MRD

Approximately 850 patients (600 cutaneous melanoma, 250 uveal melanoma) will be enrolled from 50 centres to screen for HLA-A*0201 status and then followed for up to 24 months for MRD at those same centres. Patients identified with MRD will be invited to be treated with tebentafusp at up to 10 treating centres in the UK. Patients in cohorts A and B will receive up to six months of tebentafusp, administered weekly IV, and then will be followed-up for 12 months for molecular and clinical relapse.

Patients will be in the pre-screening phase for determination of HLA-A*0201 status for up to 2 weeks. Those patients who are positive for HLA-A*0201 will be followed for MRD and will attend the clinical sites for 3 monthly testing for up to 24 months. Patients will leave the study if no molecular relapse is detected during the molecular screening period. When MRD is identified, patients will be evaluated for eligibility to enter the main study at one of up to 10 specialist treatment centres, where patients will enter the screening period for determination of eligibility to start tebentafusp administration within 6 weeks. After a maximum 6 months treatment patients will be followed up for 12 months, or until the study is completed, if this is longer.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in cohort A or B if all of the following criteria apply:

1. Uveal or cutaneous melanoma with MRD detected in molecular screening, and repeat confirmation of MRD in the sample taken as part of screening for the main study.
2. Written (signed and dated) informed consent.
3. Male or female, Age 18 years and above.
4. Life expectancy of at least 3 months.
5. ECOG performance score of 0 or 1.
6. No evidence of metastatic disease on a CT scan of neck/thorax/abdomen/pelvis for cohorts A and B and also on MRI liver for uveal melanoma for cohort B.
7. Those receiving prior immunotherapy must have recovered from any immune-mediated adverse events (≤ grade 1) other than endocrinopathies on stable replacement therapy.
8. Haematological and biochemical indices within normal ranges (refer to protocol for ranges)

Exclusion Criteria:

A patient will not be eligible for tebentafusp administration if any of the following apply:

1. Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to enrolment.
2. Uveal or cutaneous melanoma patients who present radiologically or clinically detectable disease during screening.
3. Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy before Screening is initiated
4. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
5. Any other active malignancy, with the exception of malignancies that were treated curatively and have not recurred within 2 years after completion of treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type
6. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV. This study does not require testing to confirm eligibility unless clinically indicated.
7. Clinically significant cardiac disease or impaired cardiac function (New York Heart Association grade ≥ 2), including myocardial infarction or unstable angina pectoris within 6 months of screening.
8. Active autoimmune disease or a documented history of autoimmune disease within 3 years of screening (diabetes mellitus, vitiligo, managed hypothyroidism, psoriasis and managed asthma are not exclusions).
9. Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity and any prior immunotherapy approach, 4 weeks is indicated as washout period
10. Presence of NCI CTCAE ≥ grade 2 toxicity (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥ NCI CTCAE grade 3) due to prior cancer therapy.
11. Patients currently requiring chronic, systemic corticosteroid therapy at any dose for longer than 2 weeks. Replacement treatment for pituitary or adrenal insufficiency is permitted. Local steroid therapies (e.g. otic, ophthalmic, intra-articular, or inhaled medications) are acceptable.
12. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment. Non-live vaccination (e.g. influenza) are permitted anytime during treatment.
13. Major surgery as defined by the investigator within 2 weeks of the first dose of study treatment (minimally invasive procedures such as bronchoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
14. Pregnant or lactating women, or women of childbearing potential unless effective methods of contraception are used.
15. Women of child-bearing potential who are sexually active with a non-sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during study treatment, and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician.
16. Male patients must be surgically sterile or use double barrier contraception method from enrolment through treatment and for 6 months following administration of the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Estimate the rate of molecular response (MR) to tebentafusp in each of 2 cohorts A. Cutaneous melanoma with MRD B. Uveal melanoma with MRD | ctDNA taken at baseline until end of treatment (maximum of 6 months)
  Best response to treatment, with partial molecular response (pMR) defined as a decrease in the allele frequency of the index mutation(s), and complete molecular response (cMR) as no detectable mutation(s)

SECONDARY OUTCOMES:
Efficacy of tebentafusp | ctDNA taken at baseline until end of treatment (maximum of 6 months); CT or MRI assessment as per standard of care
  Evaluate the efficacy of tebentafusp in each cohort - Relapse free survival at 12 months; duration of MR; overall survival
Safety and tolerability of tebentafusp | Up to 6 months of treatment
  Assess the safety and tolerability of tebentafusp in MRD. Incidence and severity of adverse events according to NCIC CTCAE v5.0/2019 Lee et all criteria; dose reductions, interruptions and cessations in the course of treatment
Assess the rate of molecular relapse in; A. Cutaneous melanoma B. Uveal melanoma | ctDNA taken at baseline and every 3 months during molecular screening
  Percentage of patients with molecular relapse at baseline, within 6 months and over 12 months of monitoring

OTHER OUTCOMES:
Changes in peripheral T cell populations and in serum cytokines and other analytes | Up to 6 months of treatment
  From blood drawn every 4 weeks
Preliminary evaluation of response rate in gp100 expressing melanoma | ctDNA taken at baseline until end of treatment (maximum of 6 months)
  Best molecular response in cohorts A and B

CONTACTS AND LOCATIONS:
Overall Officials: Mark Middleton, Principal Investigator — Consultant Medical Oncologist and Professor of Experimental Cancer Medicine
Locations (10):
- United Kingdom (10):
  - Cambridge University Hospitals NHS Foundation Trust (Screening only), Cambridge
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre, Liverpool
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Mount Vernon Cancer Centre, Middlesex
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Churchill Hospital, Oxford University Hospitals NHS Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust (Screening only), Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No